CLINICAL TRIAL: NCT05328089
Title: Vacuolar ATPase and Drug Resistance of High Grade Gliomas: a Study to Investigate Possible Therapeutic Roles for Proton Pump Inhibitors
Brief Title: Vacuolar ATPase and Drug Resistance of High Grade Gliomas
Acronym: GLIODRUG-V
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Principal Investigator, Carlo Giorgio Giussani, Associate Professor, University of Milano Bicocca
Other Study IDs: 0031436
Record Dates: First submitted 2022-01-15; First posted 2022-04-14 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Glioblastoma Multiforme
Keywords: V-ATPAse; Cancer Stem Cells; Glioma Metabolism
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor specimens and blood samples for patients that survives at least 12 months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
GBMs are still considered tumors with few available treatment options that are able only to achieve a temporary local control of the disease. In case of a GBM, tumor recurrence is generally expected within 12 months and it is due to the presence of marginal tumoral cells with pro-oncogenic molecular phenotypes that are resistant to actual chemotherapies and to radiation therapy. Nowadays, surgery still represent the first treatment option in case of suspected GBM and it aims to remove the contrast enhancing lesion seen at the pre-operative brain MRI. In particular, the peripheral layer of the tumor is made of low replicating cellsglioblastoma-associated stromal cell (GASC) that can show different carcinogenic properties and that are probably responsible for tumor recurrence. Metabolism of GBMs is mainly anaerobialglicolisis that leads to the transformation of glucose in ATP and lactates. The production of high lactate levels determines a decrease of intracellular pH that is counterbalanced by V-ATPase activity through H+ ions extrusion from the intracellular to the extracellular environment. Increased V-ATPase activity affects different pro-tumoral activities and plays a crucial role in chemoresistance. In fact, a low extracellular pH can reduce the efficacy of antineoplastic agents since a low pH might affect the structural integrity of drugs and their ability to pass through the plasmatic membrane. Finally, V-ATPase can act as an active pump able to excrete antineoplastic agents. GBMs with high V-ATPAse expression are able to transmit malignant features and to activate proliferation of GASC in vitro through a network of microvescicles (MV) like exosomes and large oncosomes (LO) that transport cell to cell copy DNA (cDNA) and micro-RNAs (miRNA).In this view, our work is intended to study: 1) the effects of proton pump inhibitors (PPI) on CSC and GASCs cultures as in vitro add-on treatments; 2) the MVs load (in terms of miRNAs and cDNAs) during the neuro-oncological follow-up in order to understand how it changes after surgery and adjuvant treatments; 3) the possible roles of V-ATPase as a clinical marker to be used to check tumor response to adjuvant treatments.

DETAILED DESCRIPTION:
GBMs are still considered tumors with few available treatment options that are able only to achieve a temporary local control of the disease. In case of a GBM, tumor recurrence is generally expected within 12 months and it is due to the presence of marginal tumoral cells with pro-oncogenic molecular phenotypes that are resistant to actual chemotherapies and to radiation therapy. In particular, in case of GBM it is possible to distinguish three neoplastic layers within the tumor that show different molecular patterns: the central core; the intermediate layer and the peripheral layer. Nowadays, surgery still represent the first treatment option in case of suspected GBM and it aims to remove the contrast enhancing lesion seen at the pre-operative brain MRI. In particular, the peripheral layer is made of low replicating cells and it can be considered normal when tissue sampling is made far from the tumor cavity. In fact, Clavreul et al. in 2015 demonstrated that peripheral GBM layer contains glioblastoma-associated stromal cell (GASC) that can show different carcinogenic properties and that are probably responsible for tumor recurrence. These findings can be considered in line with previous studies that showed some invasive tumor cells, various types of reactive cells, and angiogenesis with different immunophenotypes in peritumoral brain edema.

Nevertheless, some research teams are trying to understand if surgical removal of peritumoral FLAIR hyperintensity is able to reduce the tumor recurrence rate prolonging the OS.

Metabolism of GBMs is mainly anaerobial and it is sustained by glycolysis. Anaerobial glycolysis is a simple metabolic reaction that leads to the transformation of glucose in ATP and lactates. Glucose is delivered to the tumor through neoangiogenetic processes. Production of a significant amount of lactates determines a decrease of intracellular pH that is counterbalanced by V-ATPase activity through the extrusion of H+ ions from the intracellular to the extracellular environment. In vitro inhibition of V-ATPAse has proved to increase CSC apoptosis due to decrease of intracellular pH.

Moreover, increased V-ATPase activity determines an extrusion of H+ ions in the extracellular environment that can positively affect different pro-tumoral activities. In fact, a decrease of extracellular pH leads to activation of proteases able to destroy the extracellular matrix. Such activity enhances tumor spreading. Moreover, a low extracellular pH can reduce the efficacy of antineoplastic agents since a low pH might affect the structural integrity of drugs and their ability to pass through the plasmatic membrane. Finally, V-ATPase can act as an active pump able to excrete antineoplastic agents.

For this reason, PPIs are considered new anti-cancer drugs able to increase tumoral cell death, reduce tumor invasion and increase chemotherapy efficacy.

Moreover, GBMs with high V-ATPAse expression has proved to be able to transmit highly malignant features through a network of MVs and to activate proliferation of GASC in vitro through the transmission of G1 subunit of V-ATPAse.

In this view, our work is intended to study: 1) the effects of PPIs on CSC and GASCs cultures as in vitro add-on treatments; 2) the MVs load in terms of miRNAs and DNA (ssDNA, exoDNA) during the neuro-oncological follow-up in order to understand how it changes after surgery and adjuvant treatments; 3) the possible roles of V-ATPase as a clinical marker to be used to check tumor response to adjuvant treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients => 18 years old;
* Patients with an intra-axial brain tumor suspect for glioma;
* Patients able to sign a consent form for research purpose;
* Patients with planned craniotomy for brain tumor resection.

Exclusion Criteria

* Patients < 18 years old;
* Patients with known brain tumors different than gliomas;
* Patients unable to sign a consent form for research purpose;
* Patients undergoing brain tumor biopsy;
* Patients with poor intra-operative or small surgical sample for histopathological diagnosis;
* Histology diagnostic for tumors different than gliomas.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgical removal of suspect intra-axial high grade glioma and undergoing adjuvant treatments
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-01-30 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Proton Pump Inhibitors on Glioma Stem Cells | 12 months
  Testing of PPIs on cultures of Glioma Stem Cells

SECONDARY OUTCOMES:
Isolation of Exosomes from patients under neuro-oncological follow-up | 12 months
  Blood sampling of patients under neuro-oncological follow-up in order to measure the variability of exosomes and of their contents

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Socio Sanitaria Territoriale Monza - Ospedale San Gerardo, Monza, Italy

DOCUMENTS (1):
  • Study Protocol (2019-06-07): https://cdn.clinicaltrials.gov/large-docs/89/NCT05328089/Prot_000.pdf